CLINICAL TRIAL: NCT07337681
Title: Effect of a Wearable Technology-Supported Exercise Program on Fatigue and Health-Related Quality of Life in Pediatric Cancer Patients: A Randomized Controlled Trial
Brief Title: Wearable Technology-Supported Exercise Program for Fatigue and Quality of Life in Pediatric Cancer Patients (WE-EX PedsCa)
Acronym: WE-EX PedsCa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yagmur Berktas, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IU-PHO-EX-2026
Record Dates: First submitted 2026-01-04; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Cancer; Cancer-related Fatigue; Quality of Life; Exercise
Keywords: Pediatric oncology; adolescent cancer; wearable technology; exercise intervention; physical activity; cancer-related fatigue; health-related quality of life; mobile health; digital exercise program
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a single-center, parallel-group randomized controlled trial in which participants are assigned in a 1:1 ratio to either an intervention group receiving a wearable technology-supported structured exercise program or a control group receiving standard care with passive monitoring. Outcomes are assessed concurrently in both groups over an 8-week study period.
Masking Description: This is an open-label study. Due to the nature of the exercise intervention, participants and study personnel are aware of group assignment. Treating pediatric oncologists are not informed of allocation and are not involved in outcome assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wearable Technology-Supported Exercise Program (Experimental): A structured, video-guided exercise program delivered via a mobile application and supported by continuous monitoring using a wearable activity tracker.
  Interventions: Other: Wearable Technology-Supported Exercise Program
- Standard Care with Passive Monitoring (Active Comparator): Participants assigned to this arm will receive standard pediatric oncology care without a structured exercise program. Participants will wear a wearable activity tracker for passive monitoring of physical activity, heart rate, and sleep patterns only.
  Interventions: Other: standart care

INTERVENTIONS:
Other: standart care — Usual pediatric oncology care with passive wearable monitoring and no structured exercise guidance.
  Arms: Standard Care with Passive Monitoring
Other: Wearable Technology-Supported Exercise Program — Wearable Technology-Supported Exercise Program
  Arms: Wearable Technology-Supported Exercise Program

SUMMARY:
Children and adolescents receiving cancer treatment often experience fatigue, reduced physical activity, and decreased quality of life. Although exercise has been shown to reduce these problems, maintaining regular and safe physical activity during cancer treatment can be difficult due to treatment side effects, safety concerns, and limited access to supervised programs.

This study aims to evaluate the feasibility, safety, and effectiveness of a wearable technology-supported exercise program on fatigue and health-related quality of life in pediatric cancer patients aged 13 to 18 years. Participants will be randomly assigned to either an intervention group or a control group. The intervention group will participate in an 8-week structured exercise program delivered through a mobile application, including video-guided exercise sessions performed three times per week and monitored continuously using a wearable activity tracker. The control group will receive standard care and will wear the activity tracker for passive monitoring only.

Fatigue and quality of life will be assessed at baseline, mid-intervention, and after completion of the program. Physical activity, heart rate, sleep patterns, and adherence to the exercise program will be objectively monitored using wearable devices. The findings from this study are expected to provide evidence on whether a digitally delivered, wearable-supported exercise program is a feasible and beneficial approach to improving well-being in children and adolescents undergoing cancer treatment.

DETAILED DESCRIPTION:
Detailed Description

This study is a single-center, parallel-group, randomized controlled trial designed to evaluate the feasibility, safety, and efficacy of a wearable technology-supported structured exercise program on fatigue and health-related quality of life (HRQoL) in pediatric cancer patients aged 13-18 years who are receiving active cancer treatment.

Eligible participants will be randomly assigned in a 1:1 ratio to either an intervention group or a control group using stratified randomization based on age, sex, and cancer diagnosis. Allocation concealment will be ensured through a secure electronic randomization system. Treating pediatric oncologists will remain blinded to group allocation.

Study Intervention

Participants in the intervention group will take part in an 8-week structured exercise program delivered through a mobile application. The program consists of video-guided exercise sessions performed three times per week, with each session lasting approximately 40 minutes. The exercise protocol includes warm-up, aerobic, strengthening, coordination, and cool-down components and is designed to be low to moderate intensity, adaptable to individual clinical conditions, and safely performed either in seated or standing positions. Exercise content was developed by a multidisciplinary team and incorporates engagement strategies such as animated guidance and gamification elements to support adherence.

Participants in the control group will receive standard care without a structured exercise intervention. Both groups will wear a commercially available wearable activity tracker throughout the study period to allow objective monitoring of physical activity and physiological parameters. In the control group, the device will be used for passive monitoring only.

Monitoring and Assessments

Fatigue and health-related quality of life will be assessed at baseline (week 0), mid-intervention (week 4), and post-intervention (week 8) using validated, age-appropriate instruments administered through the mobile platform. Objective physical activity data, including daily step counts, active minutes, heart rate, sleep duration and patterns, and device wear time, will be continuously collected via wearable devices and securely integrated into the study database.

Functional exercise capacity will be assessed using the 6-minute walk test at the same three time points. Engagement and adherence to the intervention will be evaluated using app-based metrics such as exercise session completion, frequency of use, and participation consistency.

Safety and Feasibility

Participants will be monitored throughout the study for adverse events related to exercise participation. A pediatric hematology-oncology physician and specialist nurse will oversee clinical safety. Feasibility outcomes will include recruitment rate, retention rate, adherence to exercise sessions, and completeness of wearable-derived data.

Data Analysis

Analyses will be conducted according to the intention-to-treat principle. Changes in fatigue and HRQoL over time and between groups will be examined using appropriate repeated-measures statistical methods based on data distribution. Secondary analyses will explore changes in physical activity, sleep parameters, and engagement metrics. Effect sizes will be calculated to inform the design of future multicenter trials.

Study Purpose

This trial aims to generate preliminary evidence on the clinical applicability of integrating wearable technology-supported exercise into pediatric oncology care. The findings are intended to inform larger-scale studies and contribute to the development of scalable, evidence-based digital exercise interventions for children and adolescents undergoing cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13 to 18 years.
* Diagnosed with cancer and followed at a pediatric hematology-oncology clinic.
* Currently receiving active cancer treatment and has completed at least one cycle of chemotherapy.
* Clinically stable and medically cleared by the treating physician to participate in low-to-moderate intensity exercise.
* Able to understand instructions and communicate verbally.
* Willing to participate in at least 75% of the prescribed exercise sessions.
* Written informed consent obtained from a parent or legal guardian and assent obtained from the participant.

Exclusion Criteria:

* Presence of acute infection, uncontrolled cardiac or pulmonary disease, respiratory failure, or uncontrolled hypertension.
* Severe neurological, psychiatric, or musculoskeletal conditions that limit safe participation in exercise.
* Persistent thrombocytopenia (<10,000/µL) or known coagulation disorders.
* Uncontrolled seizure disorders.
* Central nervous system metastases.
* Any medical or psychological condition deemed by the treating physician to contraindicate exercise participation or compromise study procedures.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Cancer-Related Fatigue | Baseline (week 0), mid-intervention (week 4), and post-intervention (week 8)
  Cancer-related fatigue will be assessed using a validated multidimensional fatigue scale including physical, cognitive, and general fatigue subscales. Higher scores indicate greater fatigue severity.

SECONDARY OUTCOMES:
Health-Related Quality of Life | Baseline (week 0), mid-intervention (week 4), and post-intervention (week 8)
  Health-related quality of life will be measured using the Pediatric Quality of Life Inventory (PedsQL 4.0) Cancer Module, which assesses physical, emotional, social, and school functioning.

OTHER OUTCOMES:
Exercise Adherence | Throughout the 8-week intervention period
  Exercise adherence will be evaluated based on the proportion of prescribed exercise sessions completed by participants in the intervention group, as recorded through the mobile application and wearable activity tracker.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in this study will be shared upon reasonable request. Data will be shared only after publication of the main study results and following approval of a data-sharing request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication and ending 5 years following publication.
Access Criteria: Researchers who provide a methodologically sound proposal may request access to the data. Requests will be reviewed by the principal investigator. Data will be shared in a de-identified format to protect participant confidentiality.

REFERENCES:
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC12330123/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36980130/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32391734/